CLINICAL TRIAL: NCT04070144
Title: The First Puncture Success Rate of a Novel Injeq IQ-Tip™ System in Pediatric Lumbar Punctures
Acronym: IQ-LP-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Injeq Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IQ-LP-03
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Puncture
Keywords: Spinal puncture; Lumbar puncture
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IQ-Tip (Experimental): At most four lumbar punctures with Injeq IQ-Tip(tm) system per participant
  Interventions: Device: IQ-Tip(tm) system

INTERVENTIONS:
Device: IQ-Tip(tm) system — Physician performs therapeutic or diagnostic lumbar puncture using Injeq IQ-Tip(tm) system

SUMMARY:
The investigation aims to demonstrate the first puncture success rate, as proxy of clinical benefit and clinical performance, of bioimpedance spectroscopy based spinal needle guidance method among pediatric hemato-oncology patients requiring lumbar punctures.

DETAILED DESCRIPTION:
The primary purpose of the investigation is to demonstrate the claimed clinical benefit and safety of Injeq IQ-Tip™ system.

IQ-Tip™ is similar to common spinal needles with a custom-made stylet that enables the real-time bioimpedance measurement at the tip of the needle. The needle is connected to the analyzer device, which provides real-time CSF detection during lumbar puncture from the very tip of the needle and by these means assists conducting the medical procedure.

The investigation aims to demonstrate the first puncture success rate, as proxy of clinical benefit and clinical performance, of bioimpedance spectroscopy based spinal needle guidance method among pediatric hemato-oncology patients requiring lumbar punctures.

The investigation is conducted in the pediatric hematology and oncology units of three Finnish university hospitals

ELIGIBILITY:
Inclusion Criteria:

* Pediatric hemato-oncology patients whose diagnosis or treatment plan requires lumbar puncture to acquire a CSF sample or to inject drug or other substance
* Written and signed informed consent before the procedure from the parent and/or patient depending on the age of the patient

Exclusion Criteria:

* Parents and/or patient refusal to participate or parents and/or patient unable to give informed consent
* Any contraindications to a lumbar puncture. Contraindications include skin infection around the puncture area, unstable hemodynamics, bleeding tendency and increased intracranial pressure

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sauli Palmu, PhD MD, Principal Investigator — Tampere University Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, New Children's Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lumbar puncture
Period: Overall Study
Arm/Group | IQ-Tip
Started | 50; 152 lumbar puncture
Completed | 50; 152 lumbar puncture
Not Completed | 0; 0 lumbar puncture

BASELINE CHARACTERISTICS:
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
Age, Continuous [Mean (Full Range); unit: years] | 7.1 [1.8 to 16.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Height [Mean (Full Range); unit: cm] | 123 [85 to 178]
Weight [Mean (Full Range); unit: kg] | 29 [13 to 71]

OUTCOME MEASURES:

1. Primary Outcome: The First Puncture Success Rate
Description: Each individual lumbar puncture procedure is assessed as either 'first puncture success' or '-failure'.
  Success rate = Successes / All procedures
  Definition of the first puncture success:
  * Only one skin puncture with the needle is allowed;
  * Multiple stylet removals and reinsertions are allowed;
  * Multiple needle reorientations are allowed as long as needle tip remains inside the skin;
  * Physician must be able obtain a cerebrospinal fluid (CSF) sample that is sent to a laboratory analysis or to inject the intended medication to the patient's subarachnoid space; and
  * Physician conducting the puncture remains the same during the procedure
Time Frame: The assessment immediately following each lumbar puncture procedure
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Units Other Than Participants: Lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (Lumbar puncture) | 152
percentage of procedures | 79.5 [72.1 to 85.6]

2. Primary Outcome: Rate of Serious Adverse Events
Description: Total number of serious adverse events caused by the device. Serious adverse event in probable or causal relationship to the investigational device exposure
Time Frame: The assessment during four-week follow-up after each lumbar puncture procedure
Measure: Number; unit: SAEs
Units Other Than Participants: Lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (Lumbar puncture) | 152
SAEs | 0

3. Secondary Outcome: Percentage of Procedures With Post-dural Puncture Headache (PDPH)
Description: PDPH defined as headache that:
  * worsens in sitting or standing position
  * eases when lying down
  * occurs within 7 days after the lumbar puncture procedure
  Possible symptoms are recording using a diary filled by the patient or parents and verified by the study nurse.
Time Frame: The assessment during 7-day follow-up after each lumbar puncture procedure
Measure: Number; unit: percentage of procedures
Units Other Than Participants: Lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (Lumbar puncture) | 152
percentage of procedures | 6

4. Secondary Outcome: Percentage of CSF Samples With Greater or Equal to 10 Erythrocytes / mm^3
Description: Erythrocyte (red blood cell) count according to laboratory analysis in units of 10^6/liter or 1/mm3
Time Frame: The laboratory analysis within 3 hours of the lumbar puncture
Population: A CSF sample was successfully obtained in 150 out of 152 lumbar puncture procedures
Measure: Number (95% Confidence Interval); unit: percentage of CSF samples
Units Other Than Participants: CSF sample
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (CSF sample) | 150
percentage of CSF samples | 17.3 [11.7 to 24.4]

5. Secondary Outcome: Percentage of Procedures With Other Complications or Adverse Events
Description: E.g. PDPH or backache
  Possible symptoms are recorded using a diary filled by the patient or parents and verified by the study nurse. Diary is an open questionaire that is intended for recording any possible complication. Possible complications are not considered as pre-determined outcome measures, with the exception of Outcome #3 (rate of PDPH)
  Four-week follow up conducted by the study nurse from the hospital registers
Time Frame: The assessment during 7-day and four-week follow ups
Measure: Number; unit: percentage of procedures
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
percentage of procedures
  Nausea | 15
  Headache | 14
  Backache | 14
  Fever | 7

6. Secondary Outcome: Aggregate Sensitivity of CSF Detection
Description: The CSF detection performance of the investigational device is assessed by the physician.
  Each individual lumbar puncture procedure is classified as either 'True Positive CSF detection (TP)', 'False Negative CSF detection (FN)' or 'Procedure failed (Fail)' by the investigator.
  The aggregate sensitivity = Number of TPs / Total number of procedures
Time Frame: The assessment immediately following each lumbar puncture procedure
Measure: Number (95% Confidence Interval); unit: percentage of succesfull procedures
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
percentage of succesfull procedures | 86.1 [79.2 to 91.4]

7. Secondary Outcome: Aggregate False Detection Rate of CSF Detection
Description: Each individual lumbar puncture procedure is classified as either 'One or more False Positive CSF detections (FP)' or 'No False Positive CSF detections (TN)'.
  The aggregate false detection rate = Number of FPs / Total number of procedures
Time Frame: The assessment immediately following each lumbar puncture procedure
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
percentage of procedures | 9.2 [5.1 to 15.0]

8. Secondary Outcome: Number of Required Attempts Per Successful Lumbar Puncture Procedure
Description: In line with definition of 'the first puncture success rate', attempt is defined as: any new penetration of skin is considered a new attempt.
  Lumbar puncture is considered successful irrespective of the number of punctures if the CSF sample was eventually obtained and/or the injection of medicine could be performed
Time Frame: The assessment immediately following each lumbar puncture procedure
Measure: Mean (Full Range); unit: lumbar puncture attempt
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
lumbar puncture attempt | 1.3 [1 to 4]

9. Secondary Outcome: Number of Failed Lumbar Puncture Procedures
Description: Procedure is considered failed if physicians, even after multiple attempts, conclude that the lumbar puncture cannot be completed with available personnel or equipment due to any reason
Time Frame: The assessment immediately following each lumbar puncture procedure
Measure: Number; unit: failed procedure
Units Other Than Participants: lumbar puncture
Arm/Group | IQ-Tip
Number analyzed (Participants) | 50
Number analyzed (lumbar puncture) | 152
failed procedure | 1

ADVERSE EVENTS:
Time Frame: 4 weeks after a lumbar puncture procedure
Description: 4 week follow-up from the hospital records
Arm/Group | IQ-Tip
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 7/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQ-Tip (N=50)
Various aches (Musculoskeletal and connective tissue disorders) | 5 (5) — head, back, stomach or limbache
vomitting / nausea (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04070144/Prot_SAP_000.pdf